CLINICAL TRIAL: NCT00450567
Title: Monitoring Targeted Lung Cancer Treatments With FDG-PET/CT
Brief Title: Glucose Metabolism in Patients With Non-Small Cell Lung Cancer Treated With Targeted Therapy and Chemotherapy
Status: Completed | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000423222; P50CA086306 (NIH); UCLA-0410068-01
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-08

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: computed tomography
Procedure: positron emission tomography
Radiation: fludeoxyglucose F 18

SUMMARY:
RATIONALE: Measuring changes in glucose metabolism in patients with cancer may help doctors predict how patients respond to treatment.

PURPOSE: This clinical trial is studying glucose metabolism in patients with non-small cell lung cancer treated with targeted therapy and chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the prognostic significance of changes in glucose metabolism measured by fludeoxyglucose F 18 positron emission tomography (FDG-PET)/CT scan in patients with non-small cell lung cancer treated with targeted drugs comprising gefitinib, erlotinib hydrochloride, or other ErbB inhibitors, cyclooxygenase-2 inhibitors, or estrogen receptor blockers in combination with conventional chemotherapy.

OUTLINE: This is a prospective study.

Patients undergo fludeoxyglucose F 18 positron emission tomography (FDG-PET) scan and CT scan at baseline and at 2 weeks and 12 weeks after receiving targeted anticancer treatment. Metabolic changes detected by FDG-PET and size changes identified by CT scan are related to patient outcome and tumor response to treatment.

PROJECTED ACCRUAL: A total of 120 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer
* Any disease stage allowed
* Undergoing targeted treatment

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with non-small cell lung cancer (stage III B or stage IV) and will be treated with an experiemntal drug or a combination of chemotherapy and new drugs, as part of standarad of care or because of enrollment in a study protocol.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2004-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Correlation of glucose metabolic response with progression-free survival, overall survival, and changes in tumor size as measured by fludeoxyglucose F 18 positron emission tomography/CT scan | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Czernin, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States